CLINICAL TRIAL: NCT05100641
Title: Randomized Phase 3 Trial of Standard Care Plus AV-GBM-1 vs Autologous Monocytes as Adjunctive Therapy Following Primary Surgery Plus Concurrent Radiation-temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: AV-GBM-1 vs Control as Adjunctive Therapy Following Surgery and RT/TMZ in Newly Diagnosed GBM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aivita Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-GBM-P02-US
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Primary Glioblastoma

STUDY DESIGN:
Intervention Model Description: Double-blind, 2:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AV-GBM-1 (Experimental): Autologous dendritic cells loaded with autologous tumor antigens cryopreserved in CryoStor 5, and admixed 500 mcg GM-CSF diluted in saline
  Interventions: Biological: AV-GBM-1
- Autologous monocyte control (MC) (Placebo Comparator): Autologous monocytes cryopreserved in CryoStor 5, and admixed 500 mcg GM-CSF diluted in saline
  Interventions: Biological: Autologous monocytes

INTERVENTIONS:
Biological: AV-GBM-1 — Therapeutic autologous dendritic cell vaccine
  Arms: AV-GBM-1
Biological: Autologous monocytes — Autologous monocyte control
  Arms: Autologous monocyte control (MC)

SUMMARY:
This is a multi-center, double-blind, 2:1 randomized phase III trial to determine whether the addition of AV-GBM-1, a therapeutic, patient-specific dendritic cell vaccine, to standard therapy increases OS of patients with a recent diagnosis of primary GBM.

The intent is to enroll approximately 726 patients for tumor collection to enroll 690 who are eligible for treatment at the time of randomization and who have granted consent for participation. Because of the lack of toxicity, there are no restrictions related to performance status or blood tests at the time of treatment. The key endpoint is OS from date of first injection after RT/TMZ; secondary endpoints are PFS from date of first injection, and OS and PFS from date of randomization prior to RT/TMZ. Date of PFS will be determined by the principal investigator at each site.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, 2:1 randomized phase 3 trial to determine whether the addition of AV-GBM-1 to standard therapy increases OS of patients with a recent diagnosis of primary GBM.

Patients will sign two treatment-related consents, one for obtaining fresh tumor tissue at the time of craniotomy for the purpose of establishing a short-term tumor cell line and for awareness of subsequent leukapheresis procedure, and the other for randomization and participation in the randomized trial. As required for related medical procedures, patients will sign medical consents for craniotomy/tumor resection, and for leukapheresis to obtain monocytes for the MC control arm, or to manufacture DC.

Key eligibility criteria are (1) recovered from maximal safe surgical resection surgery from which a short-term cell culture has been established, (2) undergone leukapheresis prior to planned concurrent RT/TMZ, from which a sufficient number of MC have been derived, (3) screened, stratified and randomized prior to starting RT/TMZ. Patients will be stratified by age (70 years or greater or less than 70), KPS (90 or 100 vs 70 or 80), MGMT promotor-methylation (yes or no), and IDH-mutation status (mutated or wild-type), then randomized 2:1 (AV-GBM-1 vs MC control).

The final products will be manufactured while the patient is being treated with RT/TMZ. After recovery from RT/TMZ, one of the study agents, either the DC-ATA AV-GBM-1 or autologous MC control, will be administered weekly for three weeks just prior to starting adjuvant TMZ, and then every four weeks concurrently with, adjuvant TMZ or second-line therapy per managing physician. Both products are admixed with adjuvant 500 mcg of GM-CSF by a local pharmacist, just prior to each injection. The pharmacist, the patient, their health care givers and local research team will be masked as to whether the patient is receiving AV-GBM-1 or MC control, which are similar in appearance. Only the AIVITA manufacturing team will be aware of randomization so that the appropriate product can be manufactured per SOPs.

The first 3 weekly SC injections of study agent will be administered prior to beginning adjuvant or salvage temozolomide, temozolomide plus bevacizumab, or temozolomide plus tumor treating fields. Thereafter study agents will be injected about every 28 days for up to 18 additional vaccines (i.e. a total of 21 vaccines over 18 months from the start of investigational therapy. Depending on the number of study-agent doses available, additional leukaphereses and manufacturing of more study agent may be required if treatment is to continue up to 18 months from the start of therapy. In previous trials, 8 total injections were given over 6 months. In this trial up to 21 doses may be given over 18 months.

In previous trials each patient-specific batch of DC-ATA was divided into 10 aliquots, 8 of which were intended for injection. The range of cells was from 1 to over 30 million per aliquot. However, the clinical trials have consistently suggested that 1 to 2 million cells is a sufficient dose. Therefore, for this trial each patient-specific batch of DC-ATA will be divided into aliquots containing 2 million DC-ATA cells (prior to cryopreservation), and after the initial series of three weekly injections, subsequent injections will be administered up to 18 months from the first injection. If the product is used up, a cryopreserved cell line can be re-expanded and an additional leukapheresis procedure performed in order to make more AV-GBM-1 or MC control, if the patient and their physician wish to continue treatment. For those who were randomized to AV-GBM-1, a GBM cell culture would be re-established from a cryopreserved sample of the original cell line. If for some reason the cell line cannot be reestablished, then patients randomized to the AV-GBM-1 arm would receive injections of their monocytes with GM-CSF to preserve the double-blind conditions.

Patients who are confirmed to have experienced PD while on study must discontinue AV-GBM-1 treatment.

The intent is to enroll approximately 1,120 patients for tumor collection to have 672 patients who are eligible for treatment at the time of randomization and who have granted consent for participation. Because of the lack of toxicity, there are no restrictions related to performance status or blood tests at the time of treatment. The key endpoint is OS from date of randomization; secondary endpoints are OS and PFS from date of first injection. Date of PFS will be determined by the principal investigator at each site.

ELIGIBILITY:
Inclusion Criteria:

* For tumor collection: Age >18, Presumptive diagnosis of primary GBM with plans for surgical resection, Written informed consent to provide tumor and blood and intent to proceed with leukapheresis
* For randomization: Confirmation of GBM histology, AIVITA Biomedical confirmation of established cancer cell line and sufficient monocytes derived from PBMC during leukapheresis collection, age 70 years or greater or less than 70, KPS 90 or 100 vs 70 or 80, MGMT promotor methylation classified as positive or negative, IDH mutation classified as mutated or wild-type, and planning to initiate RT/TMZ. Written informed consent for randomization and treatment per protocol

Exclusion Criteria:

* For tumor collection: Prior history of astrocytoma or other glial tumor, Known autoimmune disease or immunodeficiency. Diagnosis of any other invasive cancer or disease process considered to be life-threatening within the next 5 years. Known allergy to GM-CSF
* For randomization: Active infection or other active medical condition that could be life-threatening, Diagnosis of underlying cardiac disease that requires active medical treatment, Pregnant, Enrolled in another investigational trial to receive an investigational treatment, KPS < 70, Did not meet inclusion/exclusion criteria for tumor collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival from date of randomization | 2.0 years
  Overall survival

SECONDARY OUTCOMES:
PFS from date of first AV-GBM-1 injection | 2.0 years
  Progression-free survival
OS from date of first AV-GBM-1 injection | 2.0 years
  Overall survival
PFS from date of randomization | 2.0 years
  Progression-free survival
Determine and compare TEAE for both study arms | 2.0 years
  Safety measurement

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Study Chair — Aivita Biomedical, Inc.

IPD SHARING:
Plan to Share IPD: No